CLINICAL TRIAL: NCT05066516
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of IN-C009 in Healthy Subjects
Brief Title: The Pharmacokinetics, Safety and Tolerability of IN-C009 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Ji-Young Park, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_DLC_101
Record Dates: First submitted 2021-09-14; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — N(beta)-fumarylcarboxyamido-2,3-diaminopropionic acid; dapagliflozin; Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1: Individual components (ICs), period 2: FCDP (Experimental): Period 1: Individual components (ICs), period 2: FCDP
  Interventions: Drug: FCDP, dapagliflozin 10mg/linagliptin 5 mg or co-administration of a single dose of dapagliflozin and linagliptin
- Period 1: FCDP, period 2: ICs (Experimental): Period 1: FCDP, period 2: ICs
  Interventions: Drug: FCDP, dapagliflozin 10mg/linagliptin 5 mg or co-administration of a single dose of dapagliflozin and linagliptin

INTERVENTIONS:
Drug: FCDP, dapagliflozin 10mg/linagliptin 5 mg or co-administration of a single dose of dapagliflozin and linagliptin — FCDP, dapagliflozin 10mg/linagliptin 5 mg or ICs, co-administration of a single dose of dapagliflozin and linagliptin

SUMMARY:
This study was conducted as a randomized, open-label, single-dose, crossover study design. All participants were randomly allocated for group A (Period 1: Individual components (ICs), period 2: FCDP) and group B (Period 1: FCDP, period 2: ICs), and each group was administered either a single dose of IN-C009 (FCDP, dapagliflozin 10mg/linagliptin 5 mg) (HK inno.N., Seoul, Korea) or co-administration of a single dose of dapagliflozin (Forxiga 10 mg, AstraZeneca, Cambridge, England, UK) and linagliptin (Trajenta 5mg, Beringer-Ingelheim, Ingelheim, Germany) after at least 10 hours of overnight fasting. After the 28 days of the washout period, the participants received the opposite treatment (Group A: IN-C009; Group B: dapagliflozin and linagliptin). The dosage of dapagliflozin and linagliptin in the study is commercially used and recommended amount for the control of T2DM currently.

On the day 1 (the day of each drug administration), the serial blood samples were drawn immediately before (0 h) and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, and 72 h (for dapagliflozin), and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, and 72 h (for linagliptin) after the each dosing to assess pharmacokinetics of each drugs.

ELIGIBILITY:
Inclusion Criteria:

* age between 19 to 45 years;
* body weight more than 50 kg

Exclusion Criteria:

* a history or evidence of hepatic, renal, gastrointestinal, or hematological abnormality;
* hepatitis B, hepatitis C, syphilis, or HIV infection;
* a history of hypersensitivity to dapagliflozin and/or linagliptin;
* clinically significant allergic disease; alcohol or drug abuse;
* heavy smoker (more than ten cigarettes per day);
* use of any medication within 30 days before the start of the study that may affect the study results.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-10-18 (Actual)

PRIMARY OUTCOMES:
Cmax | 72 hours
  peak plasma concentration
AUC | 72 hours
  area under plasma concentration versus time curve

SECONDARY OUTCOMES:
Tmax | 72 hours
  time at Cmax
half-life | 72 hours
  elimination half-life
CL | 72 hours
  clearance
Vd | 72 hours
  volume distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea